CLINICAL TRIAL: NCT04218136
Title: Cetuximab Therapeutic Drug Monitoring in Squamous Cell Carcinoma Head and Neck Cancer Patients: Determination of the Predictive Value Exposure Levels Through a Single Arm Multicentric Study
Acronym: CETUXIMAX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-36; ID RCB (Other: 2019-A02422-55)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient with head and neck cancer: Patients treated by standard treatment and have a minimum of 4 blood samples.
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples — A minimum of 4 blood samples and a maximum of 6 blood samples will be collected. Venous return blood samples collected as part of routine monitoring of patients for bioclinical parameters. Samples will be collected before start of the infusion and end of the infusion

SUMMARY:
Only about 30 percent of cancer patients have a clinical benefit upon cetuximab administration. Pilot studies in colorectal and head and neck cancer patients have suggested that cetuximab pharmacokinetics (PK), i.e. clearance values, could impact on clinical outcomes such as survival.

Determining cetuximab plasma clearance requires sophisticated PK modeling using population approaches, thus making it difficult to implement in routine clinical practice. In addition, all the preliminary studies with cetuximab were based upon Elisa determination of cetuximab plasma levels, an analytical method that fails to meet the requirements of daily practice in laboratories performing therapeutic drug monitoring. This pilot study aimed at evaluating the mass spec method analytical performance as part of a " real life " study, evaluating the inter-patient variability of exposure levels in head and neck cancer patients, and establishing a putative link between those exposure levels and clinical outcome. Results from 25 patients fully confirmed the analytical performance of the mass spec method (e.g., lack of matrix effect, acceptable sensitivity to monitor trough levels, lack of impact of sampling processing or freezing/thawing cycles). In addition, a large inter-individual variability (Superior at 50 percent) was observed, both in the peak concentrations (Cmax) and in trough levels (Cmin). Most interestingly, despite the limited number of patients enrolled, a statistically significant association was shown between exposure levels (i.e. calculated AUC) and clinical outcome (DCR). This difference was even more significant on Cmin, thus suggesting that simple trough levels monitoring could help to predict efficacy. Further analysis on survival showed that although not statistically significant, a trend towards longer both progression-free survival and overall survival was observed in the subgroup of patients with higher trough levels. In particular, 3-year survival was 29 percent and 0 percent in the subgroups with high and low trough concentrations, respectively (unpublished data).

Beyond tumoral factors, these preliminary data suggest that cetuximab Cmin levels could be a predictive marker of therapeutic efficacy and that simple therapeutic drug monitoring could help to forecast clinical outcome or enable dosage adaptation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 75 years.
* Adult patient with recurrent or metastatic histologically proven head and neck Squamous Cell Carcinoma.
* Patients to be treated by standard treatment: chemotherapy with cisplatin or carboplatin and fluorouracil in combination with a cetuximab-based protocol
* Patients having signed the non-opposition form

Exclusion Criteria:

* Patient currently participating in or having participated to a study with another investigational agent.
* Patients minor
* Pregnant or breast-feeding women.
* Any contra-indication in the Second Primary Cancers

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient with recurrent or metastatic histologically proven head and neck Squamous Cell Carcinoma. Patients will be treated by standard treatment as part of routine clinical practice
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2019-12-26 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 16 months
  Disease control rate (DCR) will be defined as the combination of complete response, partial response, and stable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Dirctor, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No